CLINICAL TRIAL: NCT01854840
Title: Betamethasone and Severity of Hyaline Membrane Disease in the Newborn Premature
Brief Title: Betamethasone and Severity of Hyaline Membrane Disease
Acronym: b-Mhyalines
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10069; 2011-A01257-34 (Other: AFSSAPS)
Record Dates: First submitted 2012-04-02; First posted 2013-05-16 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pregnant Women Receive Celesten
Keywords: hyaline membrane disease; placenta; betamethasone
MeSH Terms: conditions — Hyaline Membrane Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples will be collected. The effect of covariates as genetic polymorphism for CYP3A4, CYP3A5 and P-glycoprotein will be tested to explain the variability of placental transfer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Celesten in prevention of hyaline membrane disease.: Pregnant women that received at least a first injection of Celesten in the prevention of hyaline membrane disease.

SUMMARY:
Primary purpose: to study the relationship between betamethasone placental transfer and the occurrence and severity of the Hyaline Membrane Disease.

DETAILED DESCRIPTION:
β-Mhyalines is a prospective multicentric non interventional study. One hundred fifty pregnant women at risk of premature delivery, in the framework of Hyaline Membrane Disease of the neonate, will receive 2 intramuscular injections of Celesten (betamethasone) at 24 hours interval. Plasma samples will be collected: 2 in the mother before delivery, one maternal and one cord samples at delivery. Concentrations will be measured and analyzed using a population approach. A ratio between neonatal and maternal exposure will be calculated to represent placental transfer. The effect of covariates (genetic polymorphism for CYP3A4, CYP3A5, P-glycoprotein…, and others variables as gestational age, bodyweight at birth, apgar score, co-medication, maternal disease) will be tested to explain the variability of placental transfer. The relationship between placental transfer and the occurrence and severity of the Hyaline Membrane Disease will then be study, in order to target betamethasone maternal concentration and thus to optimize the antenatal dose to administer to the mother in the framework of Hyaline Membrane Disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who received at least a first injection of Celesten in the prevention of MMH.
* A one-term> 27 SA,
* Major Patients > or = 18 years old
* Informed Consent Form signed

Exclusion Criteria:

* Patients undergoing treatment with corticosteroids in the long term

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women (at one-term >27 PMA) that received at least a first injection of Celesten in the prevention of hyaline membrane disease
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2012-01-12 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of neonates with hyaline membrane disease | 3 days
  respiratory symptoms (respiratory rhythm disorders, signs of retraction, cyanosis, oxgen dependance >30 %). Confirmation by radiology

SECONDARY OUTCOMES:
Genetic polymorphisms | Day 1
  To study the pharmacogenetics of genetic polymorphisms that may affect the placental transfer of steroids (CYP-3A4, CYP-3A5, P-glycoprotein)
mode of delivery | Day 7
  To study the variability of the factor " mode of delivery" on fetal morbidity
blood sample of betamethasone | Day 1 and day 2
  To study the pharmacokinetics of betamethasone in all women treated
Optimal dose of betamethasone | Day 28
  Determine the optimal dose of betamethasone necessary for the prevention of MMH, especially in infants under 28 weeks
gestational age | Day 7
  To study the variability of the factors "gestational age" on fetal morbidity
birth weight | Day 7
  To study the variability of the factor " birth weight" on fetal morbidity
sex | Day 7
  To study the variability of the factor "sex" on fetal morbidity
Apgar score | Day 7
  To study the variability of the factor " Apgar score " on fetal morbidity
twinning | Day 7
  To study the variability of the factors "twinning" on fetal morbidity
time between birth and the last dose | Day 7
  To study the variability of the factor "time between birth and the last dose" on fetal morbidity
ethnicity | Day 7
  To study the variability of the factor "ethnicity" on fetal morbidity
maternal disease and treatment | Day 7
  To study the variability of the factor " maternal disease and treatment on fetal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Yves Ville, MD, PhD, Principal Investigator — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France